CLINICAL TRIAL: NCT01642563
Title: A Multi-center, Single-blind, Randomized, Parallel, Non Inferiority Study to Separately Investigate the Effect of Standard Platelets Versus Platelets Prepared With Two Commercial Procedures of Pathogen Reduction Technologies (PRT) on Bleeding Incidence and Severity in Thrombocytopenic Recipients
Brief Title: Italian Platelet Technology Assessment Study
Acronym: IPTAS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Patient enrolment below planned schedule
Sponsor: Centro Nazionale Sangue (Other Government)
Collaborators: Cerus Corporation (Industry); Terumo BCT (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ISS-2007646931
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2014-09

CONDITIONS: Leukemia; Lymphoma
Keywords: Platelet transfusion; Leukemia; Transfusion transmissible infections; Chemotherapy; Allogeneic hemopoietic stem cell transplant
MeSH Terms: conditions — Leukemia; Lymphoma | interventions — Platelet Transfusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pathogen reduced platelets (Experimental): Transfusion
  Interventions: Procedure: Platelet transfusion
- Standard platelets (Active Comparator): Transfusion
  Interventions: Procedure: Platelet transfusion

INTERVENTIONS:
Procedure: Platelet transfusion — One dose of pathogen reduced platelets
  Other Names: Intercept; Mirasol
  Arms: Pathogen reduced platelets
Procedure: Platelet transfusion — One dose of standard platelets
  Arms: Standard platelets

SUMMARY:
Italian Platelet Technology Assessment Study (IPTAS) aims at comparing bleeding frequency and severity after transfusion of standard platelets versus platelets prepared with two commercial pathogen reduction technologies (PRT) and to perform a proteomic analysis of standard versus PRT platelets. The two technologies will be analyzed separately.

Primary endpoint: incidence of bleeding of grade 2 or greater in recipients of PRT platelets versus incidence in recipients of control (standard) platelets.

Secondary endpoints: time to the first grade 2 or greater bleeding event after the first study transfusion; proportion of transfusions given to treat breakthrough bleeding; number of days with grade 2 or greater bleeding during the period of platelet transfusion support; number of platelet units transfused and total dose of platelets transfused per day of thrombocytopenic platelet support; proportion of patients with acute transfusion reactions; post-transfusion platelet count increments

Observational endpoints: frequency of human leukocyte antigen (HLA) alloimmunization, frequency of clinical refractoriness to platelet transfusion with demonstrated HLA alloimmunization, frequency of clinical refractoriness to platelet transfusion that is persistent during the period of platelet support in the absence of HLA or human platelet antigen (HPA) alloimmunization

Patients will be evaluated for 4 weeks after randomization.

DETAILED DESCRIPTION:
When patient's platelet count, done in early morning every day, falls below 10000/microliter, physician in charge issues a platelet transfusion request to transfusion service. Transfusion service (which knows patient treatment arm) issues a PRT product or a standard product as indicated, typically within hours of request receipt; patient's physician identifies unit code and intended recipient's code and determines vital signs (pulse, blood pressure, body temp). Transfusion is started and completed in 30 min. Adverse reactions are monitored by ward personnel and once a day IPTAS local coordinator visits the ward, checks IPTAS patients' records, fills IPTAS forms, examines and interviews each enrolled patient and transfers filled forms to data coordinating center in Milan.

ELIGIBILITY:
Inclusion Criteria:

1. adults (> 18 years)
2. a hematooncology diagnosis (includes patients newly diagnosed and previously diagnosed)
3. expected to require 2 or more PLT transfusions in 4 weeks
4. hospital admission (patients admitted to out-patient clinics will not be enrolled)
5. chemotherapy, related and matched unrelated donor (MUD)transplant recipients
6. recurrent auto-transplanted patients, requiring chemotherapy
7. negative pregnancy test in female patients less than 60 years old

Exclusion Criteria:

1. presence of HLA class I abs on admission with PRA >20%
2. historical documented record of 2 or more 1 hour post-TX PLT corrected count increments <5,000 per microliter
3. previously included in IPTAS
4. diagnosis of a solid tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2010-10; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence of bleeding of grade 2 or greater in recipients of PRT platelets versus incidence in recipients of control (standard) platelets | Within 4 weeks after randomization

SECONDARY OUTCOMES:
Time to the first grade 2 or greater bleeding event after the first study transfusion | Within 4 weeks after randomization
Proportion of transfusions given to treat breakthrough bleeding | Within 4 weeks after randomization
Number of days with grade 2 or greater bleeding during the period of platelet transfusion support | Within 4 weeks after randomization
Number of platelet units transfused per day of thrombocytopenic platelet support | Within 4 weeks after randomization
Proportion of patients with acute transfusion reactions | Within 4 weeks after randomization
Post-transfusion platelet count increments | Within 4 weeks after randomization
Total dose of platelets transfused per day of thrombocytopenic platelet support | Within 4 weeks after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Rebulla, MD, Principal Investigator — Fondazione Ca' Granda Ospedale Maggiore Policlinico; Stefania Frasca, Eng, Study Director — Data Management; Laura Angelici, MD, Study Director — Fondazione Ca' Granda ospedale Maggiore Policlinico
Locations (9):
- Italy (9):
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Fondazione Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Ospedale di Padova, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Policlinico Umberto I, Roma
  - Ospedale di Udine, Udine
  - Azienda Ospedaliera Verona, Verona
  - Proteomics Laboratory, Università della Tuscia, Viterbo

REFERENCES:
- [Background] Rebulla P, Grazzini G, Liumbruno GM, Aprili G, Formisano S, Girelli G, Marconi M, Salvaneschi L, Strada P, Zolla L. Pathogen inactivated platelets and prevention of immunological adverse reactions: the Italian Platelet Technology Assessment Study (IPTAS). Blood Transfus 2009;7 Suppl 1:s19-s21. DOI 10.2450/2009.0013-09.